CLINICAL TRIAL: NCT05316935
Title: Gonadotropin-releasing Hormone Agonist (GnRHa) Plus Letrozole in Non-obese Progestin-insensitive Early-stage Endometrial Cancer and Atypical Hyperplasia Patients With Conservative Treatment
Brief Title: GnRHa + Letrozole in Non-obese Progestin-insensitive Endometrial Cancer and Atypical Hyperplasia Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiaojun Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Chen, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53211030
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Neoplasms; Atypical Endometrial Hyperplasia; Progesterone Resistance
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia; Progesterone Resistance | interventions — Letrozole; Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Non-obese EEC group (G) (Experimental): 20 non-obese EEC patients will be randomized to GnRHa + Letrozole group.Then every 12 weeks, an hysteroscope will be used to evaluate the endometrial condition, and the pathological findings will be recorded.
  Interventions: Drug: GnRHa; Drug: Letrozole 2.5mg
- Non-obese EEC group (D) (Experimental): 20 non-obese EEC patients will be randomized to Diane-35 + metformin group.Then every 12 weeks, an hysteroscope will be used to evaluate the endometrial condition, and the pathological findings will be recorded.
  Interventions: Drug: Diane-35; Drug: MET
- Non-obese EAH group (G) (Experimental): 20 non-obese EAH patients will be randomized to GnRHa + Letrozole group.Then every 12 weeks, an hysteroscope will be used to evaluate the endometrial condition, and the pathological findings will be recorded.
  Interventions: Drug: GnRHa; Drug: Letrozole 2.5mg
- Non-obese EAH group (D) (Experimental): 20 non-obese EAH patients will be randomized to Diane-35 + metformin group.Then every 12 weeks, an hysteroscope will be used to evaluate the endometrial condition, and the pathological findings will be recorded.
  Interventions: Drug: Diane-35; Drug: MET

INTERVENTIONS:
Drug: GnRHa — Gonadotropin-releasing hormone analogue, intramuscular injection of 3.75mg will be given every 4 weeks , and the maximum using courses will be 6.
  Other Names: Triprorelin acetate
  Arms: Non-obese EAH group (G); Non-obese EEC group (G)
Drug: Letrozole 2.5mg — 2.5mg po qd and no more than 24 weeks
  Arms: Non-obese EAH group (G); Non-obese EEC group (G)
Drug: Diane-35 — Periodic use. Patients will receive one pill po qd for 21 days, and next period should be started after 7 days.
  Other Names: ethinylestradiol cyproterone
  Arms: Non-obese EAH group (D); Non-obese EEC group (D)
Drug: MET — 500mg po tid
  Arms: Non-obese EAH group (D); Non-obese EEC group (D)

SUMMARY:
To investigate the efficacy of GnRHa plus letrozole vs Diane-35 plus metformin in non-obese progestin-insensitive early-stage endometrial cancer (EEC) and atypical hyperplasia(EAH) patients asking for conservative treatment.

DETAILED DESCRIPTION:
There were more and more women with early endometrioid endometrial cancer (EEC) and atypical endometrial hyperplasia (EAH) who want to preserve fertility. Approximately 70% to 80% of females who meet the criteria for conservation treatment are able to achieve CR after progestin therapy, with a median time of 6-7 months, but about 20% to 30% of patients get no response or need to take longer time to achieve remission (over one year). With long duration of treatment, there will be more side effects such as weight gain, impaired liver function, endometrial injury, ovarian reserve inhibition etc. which will decrease the efficacy of conservative treatment. Previous researches had shown that GnRHa plus letrozole or ethinylestradiol cyproterone plus metformin could be a better second-line treatment for progestin-insensitive patients. Till now, no similar studies were found, so we design this study to explore the efficacy of GnRHa plus letrozole and ethinylestradiol cyproterone plus metformin in progestin-insensitive EEC and EAH patients to provide new evidences for improving conservative treatment efficacy. Considered there will be more thrombotic risks in obese patients using ethinylestradiol cyproterone, we enrolled patients with BMI < 30kg/m2 only in this study.

This will be a single-centred prospective pilot study. Patients diagnosed as progestin-insensitive EAH or EEC by dilatation and curettage (D&C) or hysteroscopy will be enrolled. Non-obese patients will be stratified by pathological diagnosis (EEC or EAH) and then they will be randomly assigned (1:1) to two arms. One will be GnRHa + letrozole group and another will be ethinylestradiol cyproterone + metformin group.

The primary endpoint is cumulative complete response (CR) rate at 28 weeks of treatment. The secondary endpoints include adverse events, duration of complete response, recurrent rate, pregnancy rate and quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed initial pathological diagnosis based upon hysteroscopy: histologically prove EAH or well-differentiated EEC G1 without myometrial invasion
* BMI<30kg/m2
* No signs of suspicious extrauterine involvement on enhanced magnetic resonance imaging (MRI) or enhanced computed tomography (CT) or ultrasound
* Using progestin, any of the following therapy, as first-line treatment:

  1. Megestrol acetate ≥ 160 mg qd using, combined with Levonorgestrel Lntrauterine System (LNG-IUS) inserted or not
  2. Medroxyprogesterone acetate ≥ 250 mg qd using, combined with LNG-IUS inserted or not
  3. LNG-IUS inserted
* Progestin-insensitive:

  1. remained with stable disease after 7 months of progestin use
  2. did not achieve CR after 10 months of progestin use
* Have a desire for remaining reproductive function or uterus
* Good compliance with adjunctive treatment and follow-up

Exclusion Criteria:

* Combined with severe medical disease or severely impaired liver and kidney function
* Pathologically confirmed as endometrial cancer with suspicious myometrial invasion or extrauterine metastasis
* Patients with other types of endometrial cancer or other malignant tumors of the reproductive system
* Patients with breast cancer or other hormone- dependent tumors or diseases that cannot be used with Diane-35, GnRHa, Letrozole or MET
* Strong request for uterine removal or other conservative treatment
* Known or suspected pregnancy
* Acute severe disease such as stroke or heart infarction or a history of thrombosis disease
* Smoker(>15 cigarettes a day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rates within 28 weeks of treatment | From date of randomization until the date of CR, assessed up to 28 weeks
  The cumulative 28-week CR rates will be calculated in two groups. Patients will be evaluated with an hysteroscopy every 12 weeks. For some may delay the evaluation as personal reasons, we define the primary outcome measure as complete response rates within 28 weeks of treatment.

SECONDARY OUTCOMES:
Adverse events | From date of randomization until the date of CR or date of hysterectomy, assessed up to 28 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be recorded, as well as incidence of adverse events.
Time to achieve complete response | From date of randomization until the date of CR or date of hysterectomy, assessed up to 28 weeks.
  The median CR time will be calculated in two groups
Relapse rates | Up to 2 years after the treatment
Rates of fertility outcomes | Up to 2 years after the treatment
  Including pregnancy and live-birth rates
Compliance | Data on treatment and hysteroscopy management will be collected, and deviations from study protocol will be recorded in writing. For example, the time of drug interruptions due to related toxicities or AEs, and delay of hysteroscopy for personal reasons.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Zhou S, Xu Z, Yang B, Guan J, Shan W, Shi Y, Chen X. Characteristics of progestin-insensitive early stage endometrial cancer and atypical hyperplasia patients receiving second-line fertility-sparing treatment. J Gynecol Oncol. 2021 Jul;32(4):e57. doi: 10.3802/jgo.2021.32.e57. PMID 34085795
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34085795/